CLINICAL TRIAL: NCT03281512
Title: Saturated Fatty Acids Intake and Mortality, Diabetes, Hypertension and Overweight in the China Health and Nutrition Survey (CHNS)
Brief Title: Saturated Fatty Acids Intake and Mortality, Diabetes, Hypertension and Overweight
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: National Institute of Health and Nutrition (Other Government)
Responsible Party: Principal Investigator, Jingjing Jiao, Associate Professor, Zhejiang University
Other Study IDs: Cohort_SFA
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Morality; Diabetes; Hypertension; Overweight
Keywords: Saturated fatty acids; CHNS
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of saturated fatty acids (SFAs) intake in the development of total death, cardiovascular diseases, diabetes, hypertension and overweight are in great controversy but evidence from large population in China is scant.The investigators aim to use the data from the China Health and Nutrition Survey to assess the long-term association of SFAs intake with total mortality, diabetes, hypertension and overweight.

DETAILED DESCRIPTION:
The role of saturated fatty acids (SFAs) intake in the development of total death, diabetes, hypertension and overweight are in great controversy but evidence from large population in China is lacking.The investigators aim to utilize the data from the China Health and Nutrition Survey. The investigators will calculate the cumulative average intake of SFAs based on 3 consecutive 24-h dietary recalls in each round.Sex-specific Cox regression models will be used to estimate the relative risk.Results from our work will be used to provide epidemiological evidence for improving recommendation on SFAs intake for Chinese in dietary guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥20 with complete data on diet and follow-up time

Exclusion Criteria:

* Cardiovascular diseases
* Diabetes (for analyses of diabetes)
* Body mass index ≥ 24 kg/㎡ (for analyses of overweight)
* Hypertension (for analyses of hypertension)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHNS is an ongoing, large-scale, household-based cohort starting in 1989. The survey used a multi-stage, random cluster process to draw a sample of 9 provinces and municipal cities, which take up about half of Chinese population.
Sampling Method: Probability Sample
Enrollment: 14383 (Actual)
Dates: Start 1989-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | From baseline until death or censoring on 31 December 2011, whichever came first, assessed up to an average of 10 years
  Incidence of all-cause death, on basis of household members' report
Diabetes | From entry into the study (baseline: 1997-2009) until 2011
  Incidence of diabetes, on basis of self-reported physician diagnosis, fasting plasma glucose ≥ 7.0 mmol/l or HbA1c ≥ 6.5%

SECONDARY OUTCOMES:
Saturated fatty acids intake | From entry into the study (baseline: 1997-2009) until 2011
  Cumulative average intake of saturated fatty acids on basis of 3 consecutive 24-h dietary recalls
Hypertension | From entry into the study (baseline: 1997-2009) until 2011
  Incidence of hypertension, on basis of self-reported physician diagnosis, systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg
Overweight | From entry into the study (baseline: 1997-2009) until 2011
  Incidence of overweight, on basis of body mass index (BMI), BMI ≥ 24 kg/㎡

REFERENCES:
- [Derived] Zhuang P, Cheng L, Wang J, Zhang Y, Jiao J. Saturated Fatty Acid Intake Is Associated with Total Mortality in a Nationwide Cohort Study. J Nutr. 2019 Jan 1;149(1):68-77. doi: 10.1093/jn/nxy237. PMID 30608597